CLINICAL TRIAL: NCT06717971
Title: Evaluating the Clinical Effectiveness of an Exergame-Based Training Program Using "WarioWare: Move It!" to Enhance Physical and Cognitive Function in Older Adults With Mild Cognitive Impairment and Dementia in Rural Long-Term Care Facilities: A Randomized Controlled Trial
Brief Title: Utilization of Exergame Programs Among Elderly Residents in Rural Nursing Care Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aoyu Li (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Aoyu Li, Clinical Professor, Tainan University of Technology
Organization: Tainan University of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TainanUT; U21A20469 (Other Grant/Funding Number: National Natural Science Foundation Collaboration)
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer's Disease
Keywords: exergame; mild cognitive impairment; dementia; long-term care facilities; multicomponent training
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The training program for the intervention group utilized the Nintendo Switch game "WarioWare: Move It,". Participants engaged with the game through Joy-Con controllers, completing rapid micro-games designed to meet specific movement-oriented objectives. The "WarioWare: Move It" training program was administered twice weekly, with each session lasting 60 minutes over 12 weeks. Each session comprised three 10-minute gaming segments, interspersed with rest periods of 1 to 5 minutes to sustain participant engagement and mitigate mental fatigue. The standard care program for the control group is grounded in routine practices of long-term care facilities, aiming to sustain and enhance the physical and mental well-being of elderly residents through structured group activities. These activities encompass tailored fitness exercises, horticultural therapy, and sedentary group engagements for older adults. The program is conducted twice a week, with each session lasting 60 minutes over 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: Because of the design of the study and the nature of the interventions, blinding the staff and participants of the LTCFs is impossible. The assessors, measuring the outcomes, and the interpreter, analyzing the data, will be blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention in this group is exergame-based multicomponent training program.
  Interventions: Other: Exergame-based multicomponent training program.
- Control group (Sham Comparator): The control group received routine care in a long-term care center.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Exergame-based multicomponent training program. — The training program for the intervention group utilized the Nintendo Switch game "WarioWare: Move It,". Participants engaged with the game through Joy-Con controllers, completing rapid micro-games designed to meet specific movement-oriented objectives. Each game session lasted approximately five seconds, requiring participants to quickly adapt to various physical actions and postures, such as waving, jumping, swinging arms, rotating, and mimicking object movements. The game's dynamic structure provides an engaging experience that promotes physical coordination, reaction speed, upper and lower limb strength, and hand-eye coordination through diverse movement patterns. Switching between tasks compels players to adjust to varying motion demands swiftly, enhancing physical agility while strengthening attention-shifting and quick decision-making skills.
  Arms: Intervention group
Other: Standard care — The standard care program for the control group is grounded in routine practices of long-term care facilities, aiming to sustain and enhance the physical and mental well-being of elderly residents through structured group activities. These activities encompass tailored fitness exercises, horticultural therapy, and sedentary group engagements for older adults. The fitness exercises are adapted to meet the varying physical conditions of participants, ensuring a safe and comfortable environment that promotes moderate physical activity. Horticultural therapy involves hands-on planting and tending to plants, stimulating the senses, and fostering emotional regulation, contributing to improved psychological health. Sedentary activities, such as tabletop games, emphasize social interaction and cognitive maintenance by promoting a relaxed social environment that helps participants remain cognitively engaged.
  Arms: Control group

SUMMARY:
Background: Cognitive impairment is prevalent among older adults and frequently misdiagnosed or diagnosed late, increasingly drawing attention as a significant health issue in aging populations. Compared to community-dwelling individuals, cognitive impairments are more common among residents of long-term care facilities (LTCFs). These facilities face challenges implementing organized exercise programs due to a shortage of professional caregivers and limited resources. Additionally, older adults may lose interest in repetitive interventions over time. "WarioWare: Move It!" by Nintendo, a novel exergame that combines aerobic exercise, body coordination, balance training, and cognitive tasks, provides an immersive experience to enhance motivation and reduce staff intervention, presenting a potential solution.

Methods: The randomized controlled trial was conducted across multiple rural LTCFs in Shanxi Province, involving participants aged 65 and older. Participants were randomly assigned to either the intervention group (receiving the "WarioWare: Move It!" intervention) or the control group (receiving standard care). The intervention involved motion-sensing actions and postures (such as waving, jumping, arm swinging, rotating, and mimicking object movements) using the Joy-Con controllers for 60 minutes twice a week over 12 weeks. Primary outcome measures were derived from a battery of clinical tests, including the Sit and Reach test (the distance between the hands and toes when reaching forward), Shoulder Flexibility test (the distance between hands clasped behind the back), Trunk Rotation Flexibility test (the angle of the waist rotation to each side), Shoulder Range of Motion test (the angles of shoulder flexion, extension, abduction, and adduction), Elbow Range of Motion test (the angle of elbow flexion), Figure-of-Eight Walk test (completion time), Standing Balance test (balance duration), Hand Dexterity test (the number of blocks moved by the dominant hand in one minute), and Cognitive Function tests (e.g., Cognitive Abilities Screening Instrument, the Chinese version of the Mini-Mental State Examination, and the Montreal Cognitive Assessment). Statistical analysis was performed using mixed ANOVA, with time as the within-subject factor and intervention group as the between-subject factor, to assess the training effects on the various outcome measures.

Anticipated benefits: The intervention involving *WarioWare: Move It!* holds promise for enhancing physical flexibility, joint mobility, motor coordination, hand dexterity, and cognitive function among elderly individuals with mild cognitive impairment or dementia residing in rural care centers. This innovative and practical approach offers a viable solution for promoting health among older adults in resource-limited settings, demonstrating significant potential for broader application in similar environments.

DETAILED DESCRIPTION:
Background:

Cognitive impairment is prevalent among older adults and frequently misdiagnosed or diagnosed late, increasingly drawing attention as a significant health issue in aging populations. Compared to community-dwelling individuals, cognitive impairments are more common among residents of long-term care facilities (LTCFs). These facilities face challenges implementing organized exercise programs due to a shortage of professional caregivers and limited resources. Additionally, older adults may lose interest in repetitive interventions over time.

Despite the demonstrated clinical benefits of exergames for community-dwelling older adults, their effectiveness within LTCFs remains insufficiently explored. Current research primarily focuses on improvements in health-related quality of life, cognitive function, and overall functional status, with relatively few assessments targeting specific physical functions, such as flexibility, joint mobility, motor coordination, and hand dexterity. However, these physical capabilities are crucial for the independence of older adults. For instance, limited flexibility can hinder daily activities, directly impacting self-care abilities and increasing dependency on others. A reduction in joint mobility is often associated with joint stiffness and pain, restricting the range of motion and diminishing overall physical function, limiting the living space and activity radius of elderly individuals. Motor coordination is critical in balance maintenance and complex movements, where diminished coordination heightens the risk of falls. Falls can have severe consequences for older adults, including fractures, prolonged immobility, or even accelerated frailty, substantially reducing the quality of life. Hand dexterity also underpins the self-sufficiency of older adults. Loss of fine motor skills, such as gripping, pinching, and writing, can restrict their ability to perform daily tasks and participate socially, potentially leading to psychological distress.

The Nintendo exergame "WarioWare: Move It!" integrates twelve distinct movement modes, offering not only aerobic, coordination, and balance training but also cognitive exercises that engage memory, attention, and logical reasoning. The game's difficulty can be flexibly adjusted to match users' needs, ensuring optimal training effects at appropriate challenge levels. Despite its evident potential, comprehensive empirical studies are still required to substantiate its benefits fully. Therefore, this study conducted a 12-week longitudinal user study to examine the feasibility and potential clinical utility of "WarioWare: Move It!" for elderly populations in rural LTCFs. Furthermore, this research provides valuable insights and references for geriatric rehabilitation professionals and human-computer interaction researchers interested in designing exergame-based interventions for elderly care.

Methods:

The randomized controlled trial was conducted across multiple rural LTCFs in Shanxi Province, involving participants aged 65 and older. Participants were randomly assigned to either the intervention group (receiving the "WarioWare: Move It!" intervention) or the control group (receiving standard care). The intervention involved motion-sensing actions and postures (such as waving, jumping, arm swinging, rotating, and mimicking object movements) using the Joy-Con controllers for 60 minutes twice a week over 12 weeks. Primary outcome measures were derived from a battery of clinical tests, including the Sit and Reach test (the distance between the hands and toes when reaching forward), Shoulder Flexibility test (the distance between hands clasped behind the back), Trunk Rotation Flexibility test (the angle of the waist rotation to each side), Shoulder Range of Motion test (the angles of shoulder flexion, extension, abduction, and adduction), Elbow Range of Motion test (the angle of elbow flexion), Figure-of-Eight Walk test (completion time), Standing Balance test (balance duration), Hand Dexterity test (the number of blocks moved by the dominant hand in one minute), and Cognitive Function tests (e.g., Cognitive Abilities Screening Instrument, the Chinese version of the Mini-Mental State Examination, and the Montreal Cognitive Assessment). Statistical analysis was performed using mixed ANOVA, with time as the within-subject factor and intervention group as the between-subject factor, to assess the training effects on the various outcome measures.

Study Procedure:

Participants meeting the inclusion criteria will be recruited from long-term care facilities in Shanxi Province, including daycare centers and nursing homes. A purposive sampling method will be employed for participant selection, with the entire recruitment process strictly supervised by experienced neurologists.

Participants will be randomly assigned to either the intervention group or the control group.

All outcome measures will be assessed at baseline, after 12 weeks of intervention, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. normal or corrected-to-normal hearing and vision;
2. age over 65;
3. residence in a senior care facility or a minimum stay of one month in such a facility;
4. completion of the Global Deterioration Scale (GDS), the Chinese version of the Mini-Mental State Examination (MMSE), and the Chinese version of the Montreal Cognitive Assessment (MoCA), with the capacity to communicate effectively;
5. ability to engage in moderate physical activity without physical disability;
6. absence of severe depressive symptoms or other neurological disorders (e.g., stroke, dizziness, epilepsy);
7. provision of informed consent by the participant or their guardian.

Exclusion Criteria:

1. Individuals who have significant cardiopulmonary diseases;
2. those regularly receiving oxygen supplementation
3. those who have uncontrollable hypertension
4. those who had a recent infection or fracture or were diagnosed with other diseases that might prohibit them from participating in exercises according to the guidelines of the American College of Sports Medicine.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Sit and Reach test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The Sit and Reach test measures the participant's ability to stretch forward while seated with legs extended and heels fixed. The farthest distance reached with outstretched hands toward the toes is recorded, with the gap between the fingertips and toes serving as the flexibility index.
Shoulder Flexibility test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The Shoulder Flexibility test assesses flexibility by measuring the distance between the hands when clasped behind the back [31-32]. Participants with higher flexibility achieve either easy hand clasping or shorter hand-to-hand distance.
Trunk Rotation Flexibility test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The Trunk Rotation Flexibility test requires participants to stand with feet together, and arms extended forward, rotating the torso left and right around the waist. The maximum angle reached on each side indicates flexibility, with more prominent angles signifying greater flexibility.
Shoulder range of motion test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The participant stands upright, and the maximum range of motion of the shoulder joint is measured in the following directions: flexion, extension, abduction, and adduction.
Elbow range of motion test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The participant stands upright, and the flexion angle of the elbow joint is measured.
Figure of eight walk test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The participant walks around two markers placed on the floor in a figure-of-eight pattern, with a total walking distance of 10 meters. The time taken to complete the walk is recorded.
Standing balance test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The participant stands with their feet together and eyes closed to maintain balance. The duration for which the participant can maintain balance is recorded.
Box and block test | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The number of blocks the participants transferred in 60 seconds from one compartment to the other compartment of the wooden box.
Cognitive abilities screening instrument | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The scale is commonly used to assess mild cognitive impairment and early-stage dementia, comprising nine sections that evaluate domains such as attention, memory, orientation, language, abstract thinking, and calculation. The assessment typically takes 20 minutes to complete. Scores range from 0 to 100, with higher scores indicating better cognitive function.
Chinese version of the mini-mental state examination scale | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The scale is widely used in clinical and research settings to evaluate cognitive status through a brief question-and-answer format. It covers dimensions such as orientation, memory, attention, language skills, and visuospatial abilities. The scoring range is 0 to 30, with higher scores indicating superior cognitive performance.
Chinese version of the montreal cognitive assessment scale | The initial assessment occurred at baseline prior to randomization. Subsequent evaluations were conducted at the end of 12 weeks (post-test) and six months after the intervention concluded (after 6 months).
  The scale is a comprehensive assessment tool for cognitive performance across multiple domains. It consists of 30 items and evaluates visuospatial abilities, memory, language, calculation, abstract reasoning, attention, and orientation. The test typically takes around 10 minutes to administer. Scores range from 0 to 30, with higher scores correlating with better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Provincial People's Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
Information about the Shared Individual Participant Data (IPD) program can be obtained by contacting the registrant.

REFERENCES:
- [Result] Schattin A, Pickles J, Flagmeier D, Scharer B, Riederer Y, Niedecken S, Villiger S, Jurt R, Kind N, Scott SN, Stettler C, Martin-Niedecken AL. Development of a Novel Home-Based Exergame With On-Body Feedback: Usability Study. JMIR Serious Games. 2022 Dec 6;10(4):e38703. doi: 10.2196/38703. PMID 36472900
- [Result] Yu J, Li J, Huang X. The Beijing version of the Montreal Cognitive Assessment as a brief screening tool for mild cognitive impairment: a community-based study. BMC Psychiatry. 2012 Sep 25;12:156. doi: 10.1186/1471-244X-12-156. PMID 23009126
- [Result] Wong SS, Yam MS, Ng SS. The Figure-of-Eight Walk test: reliability and associations with stroke-specific impairments. Disabil Rehabil. 2013;35(22):1896-902. doi: 10.3109/09638288.2013.766274. Epub 2013 Apr 19. PMID 23600714
- [Result] Wang RY, Huang YC, Zhou JH, Cheng SJ, Yang YR. Effects of Exergame-Based Dual-Task Training on Executive Function and Dual-Task Performance in Community-Dwelling Older People: A Randomized-Controlled Trial. Games Health J. 2021 Oct;10(5):347-354. doi: 10.1089/g4h.2021.0057. Epub 2021 Sep 1. PMID 34491113
- [Result] Chu CH, Biss RK, Cooper L, Quan AML, Matulis H. Exergaming Platform for Older Adults Residing in Long-Term Care Homes: User-Centered Design, Development, and Usability Study. JMIR Serious Games. 2021 Mar 9;9(1):e22370. doi: 10.2196/22370. PMID 33687337
- [Result] Chen KM, Li CH, Huang HT, Cheng YY. Feasible modalities and long-term effects of elastic band exercises in nursing home older adults in wheelchairs: A cluster randomized controlled trial. Int J Nurs Stud. 2016 Mar;55:4-14. doi: 10.1016/j.ijnurstu.2015.11.004. Epub 2015 Nov 28. PMID 26655368
- [Result] Meekes W, Stanmore EK. Motivational Determinants of Exergame Participation for Older People in Assisted Living Facilities: Mixed-Methods Study. J Med Internet Res. 2017 Jul 6;19(7):e238. doi: 10.2196/jmir.6841. PMID 28684385
- [Derived] Li A, Qiang W, Li J, Geng Y, Qiang Y, Zhao J. Effectiveness of an exergame-based training program on physical and cognitive function in older adults with cognitive impairment: a randomized controlled trial in rural China. BMC Geriatr. 2025 Nov 11;25(1):892. doi: 10.1186/s12877-025-06341-6. PMID 41219720
- [Derived] Li A, Qiang W, Li J, Geng Y, Qiang Y, Zhao J. Retracted: Evaluating the Clinical Efficacy of an Exergame-Based Training Program for Enhancing Physical and Cognitive Functions in Older Adults With Mild Cognitive Impairment and Dementia Residing in Rural Long-Term Care Facilities: Randomized Controlled Trial. J Med Internet Res. 2025 Feb 19;27:e69109. doi: 10.2196/69109. PMID 39969990